CLINICAL TRIAL: NCT06750497
Title: The Impact of Short-term Forearm Immobilization on Forearm Muscle Glucose and Amino Acid Metabolism of Volunteers With or Without Type 2 Diabetes
Brief Title: Forearm Immobilization in T2D
Acronym: FIT2D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Marlou Dirks, Assistant Professor, Wageningen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NL87404.028.24
Record Dates: First submitted 2024-11-22; First posted 2024-12-27 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants with Type 2 Diabetes (Experimental): Two days of standardized meal consumption
  Interventions: Behavioral: Forearm immobilization
- Participants without Type 2 Diabetes (Experimental): Two days of standardized meal consumption
  Interventions: Behavioral: Forearm immobilization

INTERVENTIONS:
Behavioral: Forearm immobilization — Two days of forearm immobilization

SUMMARY:
The aim of the present study is to assess the impact of short-term forearm immobilization on forearm muscle glucose uptake and amino acid net balance and kinetics in individuals with T2D compared with a control group with normoglycaemia.

DETAILED DESCRIPTION:
Participants with and without T2D will undergo 2 days of forearm immobilization as a model of local physical inactivity. Before, throughout, and after immobilization arteriovenous forearm balance measurements will be combined with a stable isotope tracer infusion to measure muscle glucose uptake and amino acid balance, uptake, and efflux.

ELIGIBILITY:
Inclusion criteria

* Males and females with or without diagnosed type 2 diabetes
* Use lifestyle changes, metformin, gliclazide, or a combination thereof as oral glucose-lowering treatments for T2D
* Aged 18-80 years at the time of signing informed consent
* 18.5 ≥ BMI ≤ 35 kg·m2

Exclusion criteria

* Type 1 or a genetic form of diabetes
* Any diagnosed cardiovascular (heart) disease or high blood pressure (≥160 mmHg systolic and/or ≥100 mmHg diastolic)
* Chronic use of any prescribed or over-the-counter pharmaceuticals (excluding oral contraceptives and contraceptive devices) that interact with muscle substrate metabolism (e.g. selective serotonin reuptake inhibitors)
* Consumption of a low-carbohydrate diet
* Smoking or chewing tobacco
* Known anaemia
* Regular use of dietary protein and/or amino acid supplements (>3 times per week)
* Currently involved in a structured progressive resistance training program (>3 times per week)
* A personal or family history of thrombosis (clots)
* Any previous motor disorders or inborn errors in muscle and/or lipid metabolism
* History of kidney disease
* History of liver disease
* Pregnant or breastfeeding
* History of any drug or alcohol abuse in the past two years
* Claustrophobia
* Unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in forearm muscle glucose uptake | From 0 to 48 hours
  The change in postprandial muscle insulin sensitivity, measured as forearm glucose uptake, from pre-immobilization to post-immobilization

SECONDARY OUTCOMES:
Temporal change in forearm glucose uptake | Prior to and for 3.5 hours following every meal consumption during the 48 hours forearm immobilization period
  The change in postprandial muscle insulin sensitivity, measured as the temporal response of forearm glucose uptake (FGU), in response to repeated meals during 48 hours of forearm immobilization
Change in forearm muscle amino acid kinetics | Baseline and at regular intervals for 3.5 hours following the first and last meal consumption during the test period (0 to 48 hours)
  Plasma phenylalanine kinetics assessed using a stable isotope tracer infusion. Measurements include the rate of appearance (Ra) of phenylalanine across the forearm.
Change in forearm muscle amino acid kinetics | Baseline and at regular intervals for 3.5 hours following the first and last meal consumption during the test period (0 to 48 hours)
  Plasma phenylalanine kinetics assessed using a stable isotope tracer infusion. Measurements include the rate of disappearance (Rd) of phenylalanine across the forearm.
Change in forearm muscle amino acid kinetics | Baseline and at regular intervals for 3.5 hours following the first and last meal consumption during the test period (0 to 48 hours)
  Plasma phenylalanine kinetics assessed using a stable isotope tracer infusion. Measurements include the net balance (NB) of phenylalanine across the forearm.
Change in whole-body substrate oxidation | Measurements will be performed at baseline, and at postprandial intervals (at 1 hour, 2 hours, 3 hours) during a 0 to 48-hour test period.
  Change in whole-body substrate oxidation measured using indirect calorimetry, measured before and in response to repeated mixed meals

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University and Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No